CLINICAL TRIAL: NCT02548299
Title: Cooking and Nutrition Education for Health Among Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: The Honor Project Trust (Unknown)
Responsible Party: Principal Investigator, Linda Libertini, Research Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-1607
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Diabetes
Keywords: Diabetes; Cooking; Nutrition; Lifestyle Medicine
MeSH Terms: conditions — Diabetes Mellitus | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cooking Lecture (Experimental): Participants in this arm will receive cooking education through lecture/PowerPoint presentation led by our executive chef. Participants will also attend nutrition education classes led by our registered dietician. Lastly, e-coaching with a certified health coach will be offered to participants with access to a personal email account.
  Interventions: Other: Nutrition Education; Other: Cooking Lecture; Other: e-Coaching
- Cooking Demo (Experimental): Participants in this arm will receive cooking education through observation of our executive chef who will explain cooking techniques and healthy food preparation practices as he cooks a healthy recipe(s) for participants to sample. Participants will also attend nutrition education classes led by our registered dietician. Lastly, e-coaching with a certified health coach will be offered to participants with access to a personal email account.
  Interventions: Other: Nutrition Education; Other: Cooking Demo; Other: e-Coaching
- Hands-on Cooking (Experimental): Participants in this arm will receive cooking education through hands on practical experience with our executive chef in a teaching kitchen. Participants will be able to sample what they prepare. Participants will also attend nutrition education classes led by our registered dietician. Lastly, e-coaching with a certified health coach will be offered to participants with access to a personal email account.
  Interventions: Other: Nutrition Education; Other: Hands-on Cooking; Other: e-Coaching

INTERVENTIONS:
Other: Nutrition Education — Nutrition classes will be led by a registered dietician.
Other: Cooking Lecture
  Arms: Cooking Lecture
Other: Cooking Demo
  Arms: Cooking Demo
Other: Hands-on Cooking
  Arms: Hands-on Cooking
Other: e-Coaching

SUMMARY:
This study is a multi-dimensional therapeutic lifestyle program that offers cooking and nutrition education as well as email-based health coaching to diabetic patients in an underserved Cleveland community. This is an innovative project as it is one of the first focused efforts within this community to improve diabetes control and prevent diabetes progression through cooking and nutrition as well as to systematically measure both clinical and behavioral outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Current State of Ohio Medicaid recipient
* Current diagnosis of diabetes, as reported in the electronic medical record
* Completed at least one diabetes education visit at STJHC
* Have daily access to a functional kitchen in home

Exclusion Criteria:

* Pregnancy or lactation or plans to be pregnant or lactate during study
* Current alcoholism or abuse of recreational drugs
* Self-reported or history of HIV or hepatitis or active tuberculosis
* Travel plans that do not permit full participation especially during the first 8 study visits
* Recent unexplained weight loss (10 pounds or more in past 3 months)
* Any diagnosis that would interfere with or prevent a change in diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Investigator-Designed Cooking Skills Questionnaire - Change from Baseline to 8 weeks | 8 weeks
  Responses to individual questions will be tracked throughout the intervention in order to evaluate basic cooking skills and knowledge of nutrition that can be used to prepare healthy meals and follow recipes.
Investigator-Designed Cooking Skills Questionnaire - Change from Baseline to 6 months | 6 months
  Responses to individual questions will be tracked throughout the intervention in order to evaluate basic cooking skills and knowledge of nutrition that can be used to prepare healthy meals and follow recipes.

SECONDARY OUTCOMES:
Height (centimeters) - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Height (centimeters) - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Weight (kilograms) - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Weight (kilograms) - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Fasting Blood Glucose (mg/dL) - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Fasting Blood Glucose (mg/dL) - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Blood Pressure - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Blood Pressure - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Total Cholesterol (mg/dL) - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Total Cholesterol (mg/dL) - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
LDL Cholesterol (mg/dL) - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
LDL Cholesterol (mg/dL) - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
HDL Cholesterol (mg/dL) - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
HDL Cholesterol (mg/dL) - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Triglycerides (mg/dL) - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Triglycerides (mg/dL) - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Hemoglobin A1c (%) - Change from Baseline to 8 weeks | 8 weeks
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Hemoglobin A1c (%) - Change from Baseline to 6 months | 6 months
  Each participant's height, weight, fasting glucose, blood pressure, blood lipids (total cholesterol, LDL, HDL, triglycerides), and HgbA1c will be abstracted from their electronic medical record at baseline, 8 weeks and 6 months (+/- 2 weeks) to record changes in values.
Dietary Fat Consumption Questionnaire - Change from Baseline to 8 weeks | 8 weeks
  Questionnaire will be given at baseline, 8 weeks and 6 months to assess nutritional consumption of fat. This Block Dietary Data Screener is a validated questionnaire with scoring to show changes over the time of the program.
Dietary Fat Consumption Questionnaire - Change from Baseline to 6 months | 6 months
  Questionnaire will be given at baseline, 8 weeks and 6 months to assess nutritional consumption of fat. This Block Dietary Data Screener is a validated questionnaire with scoring to show changes over the time of the program.
Dietary Fiber, Fruit and Vegetable Consumption Questionnaire - Change from Baseline to 8 weeks | 8 weeks
  Questionnaire will be given at baseline, 8 weeks and 6 months to assess nutritional consumption of fiber, fruits and vegetables. This Block Dietary Data Screener is a validated questionnaire generating a single composite score to show changes over the time of the program
Dietary Fiber, Fruit and Vegetable Consumption Questionnaire - Change from Baseline to 6 months | 6 months
  Questionnaire will be given at baseline, 8 weeks and 6 months to assess nutritional consumption of fiber, fruits and vegetables. This Block Dietary Data Screener is a validated questionnaire generating a single composite score to show changes over the time of the program

CONTACTS AND LOCATIONS:
Overall Officials: Mladen Golubic, MD, PhD, Principal Investigator — The Cleveland Clinic